CLINICAL TRIAL: NCT03233425
Title: Evaluation of Therapy for Overweight Children and Adolescents in Switzerland: Therapy in Multiprofessional Group Programs - Part 2, Collection and Analysis of Data
Brief Title: Evaluation of Multiprofessional Group Programs for Paediatric Obesity Therapy
Acronym: KIDSSTEP
Status: Completed | Type: Observational
Sponsor: Ostschweizer Kinderspital (Other)
Collaborators: University Hospital, Geneva (Other); akj, Fachverband Adipositas im Kindes- und Jugendalter, Switzerland (Unknown); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Principal Investigator, Dagmar l'Allemand, Prof. Dr. med., Ostschweizer Kinderspital
Other Study IDs: EKSG 08/023; 09.004211/204.0001/-629 (Other Grant/Funding Number: FOPH, CH (www.aramis.admin.ch)); l'Allemand, 20110901 (Other Grant/Funding Number: Wyeth Stiftung, Zug)
Record Dates: First submitted 2015-03-04; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Overweight
Keywords: Child; adolescent; co-morbidity; psychology; motivation; physical activity; eating disorders; quality of life; therapy; predictors
MeSH Terms: conditions — Overweight; Motor Activity; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: multiprofessional group therapy — Behavioural therapy of lifestyle including activity, family and eating habits

SUMMARY:
The aim of this pilot project is to disseminate multiprofessional group programs (*MGP*) for therapy of the estimated 119'140 overweight/obese children in Switzerland. Family-based behavioral MGPs have been implemented from 2009 to 2013 to determine changes of health and family behaviours, after the intensive phase (*T1*), at 1 and 2 years after start (*T2*, *T3*). MGP costs are reimbursed in Switzerland: 1) if 116 sessions are provided by experts in physical activity, nutrition and psychology; 2) if parents are included and if their adherence is higher than 85%. In the nationwide "Evaluation of Multiprofessional Group Programs for Paediatric Obesity Therapy" (*KIDSSTEP*) study, multiple psychosocial and physical parameters were assessed at T0, T2 and T3 . Out of 33 certified centers, 25 were active and only 19 were re-certified in 2013/2014. Obese children suffer from major co-morbidities and therefore, only one third of referred patients can be treated in MGPs and their beneficial effects on obesity as well as physical and mental health outcomes are sustained over 2 years.

DETAILED DESCRIPTION:
In Switzerland, the number of overweight children <18 years is estimated to 80'000 and related cardiovascular, osteoarticular and other complications are already present in approximately in 50% of these youth. Controlled studies demonstrated that multiprofessional treatment programs can reduce adiposity and improve health risk factors. To pre-empt the deterioration of obesity and co-morbidities in adult life, the Swiss Department of the Interior (EDI) approved in 2007 the reimbursement of treatment of overweight children by health insurances , if conducted in certified multi-professional family-based group programs. All programs have to participate in a scientific evaluation study supported by the Federal Office of Public Health (FOPH) in order to determine nationwide outcomes in clinical practice. The goal of this study is to evaluate individual changes of physical activity, nutrition, behaviours, quality of life, co-morbidities and adiposity during therapy and to identify predictors of positive or negative changes.

During 5 years, the investigators will recruit about 200 children and adolescents aged 6 to 18 years every year. Patients must have a Body Mass Index (BMI), fat mass or waist circumference above the 97th percentile, or a BMI above the 90th percentile plus a co-morbidity. Together with their parents they will be enrolled in an intensive group therapy program for 6 to 12 months, with 12 months of follow up. To date, in 25 certified centres, physicians, nutrition and physical activity specialists as well as psychologists can provide a multiprofessional standardized care, the costs of participation being reimbursed after regular presence. At start, after 1 year and 2 years, standardized instruments validated in Swiss or European children will be used to document changes during therapy. Questionnaires will assess motivation, weight of parents, personal and family history, quality of life, child and family lifestyle, parenting skills, eating or psychological disorders, and satisfaction. Other investigations will include medical examination, blood tests, and European Fitness (*Eurofit*)-test for physical fitness and capacities. Anonymised data will be recorded centrally in an electronic database, after controlling for completeness and plausibility. Informed consent and positive votes of local ethical committees will be obtained. Reports on cross-sectional and longitudinal descriptive statistics and benchmarking will be provided once yearly. A comprehensive multivariate analysis of complex associations between predictors and health-related outcomes will be completed. Statistical analyses will be performed by specialists in each field and will be supervised by public health scientists. To guarantee meaningful analyses, the last patients will be included in December 2013.

ELIGIBILITY:
Inclusion Criteria:

* BMI above the 97th percentile, or in second line waist circumference or fat mass above the nor-mal range, or BMI above the 90th percentile associated with the presence of co-morbidities
* Medical examination is a pre-requisite
* Motivation of the patient and support by the family are pre-requisites
* Psychiatric diseases or severe psychosocial restraints must be adequately tackled.
* Informed consent of patients and parents to the participation in an anonymous evaluation,

Exclusion Criteria:

* healthy child
* no motivation for therapy, as assessed by interview and questionnaires to Patient and Family
* psychiatric disease without adequate treatment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Overweight children < 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 1152 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Body mass index - standard deviation score (*SDS*), (*BMI-SDS*) | 2 years
  Age- and sex-adjusted BMI according to World Health Organisation (*WHO*) charts used in Switzerland

SECONDARY OUTCOMES:
Quality of life as assessed by Quality of life questionnaires for children and adolescents (*KIDSSCREEN*) with 52 questions | 2 years
  Outcome Measure is a Scale
Eurofit - Test | 2 years
  Outcome measure is a score on physical fitness and sport activity of children and adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar lAllemand, Pr, Principal Investigator — Ostschweizer Kinderspital, St. Gallen, Switzerland
Locations (1):
- Ostschweizer Kinderspital, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No